CLINICAL TRIAL: NCT06880380
Title: The Efficacy and Safety Study of CAR-T Cells for Functional Cure in HIV-1/AIDS Patients
Acronym: HIV-CAR-T
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024087
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: HIV Infected Individuals; HIV
Keywords: CAR-T; HIV; Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental)
  Interventions: Biological: HIV-CAR-T

INTERVENTIONS:
Biological: HIV-CAR-T — Intravenous Infusion of CAR-T Cells

SUMMARY:
Autologous CAR-T cell therapy in HIV-1/AIDS patients

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years;
2. Confirmed diagnosis of HIV-1 infection, with regular antiviral therapy ≥24 months prior to enrollment and sustained HIV-RNA levels <50 copies/mL for the 12 months preceding enrollment;
3. CD4+ T-cell count >350/μl within 30 days prior to enrollment;
4. Female participants of childbearing potential (including those ≤50 years old who are amenorrheic) must have a negative urine pregnancy test; from the screening period until the end of the study, participants should have no plans for conception and must voluntarily adopt effective contraceptive measures;
5. Willingness to provide true identity information and comply with follow-up requirements;
6. Ability to fully understand the study objectives, procedures, and potential risks, voluntary signing of an informed consent form, and adherence to the study requirements.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or of childbearing potential unwilling/unable to use effective contraception.
2. Coinfection with other viruses or infections, including HIV-2, HAV, HBV, HCV, HDV, HEV, EBV, CMV, or syphilis.
3. History of AIDS-related opportunistic infections or malignancies within the past year (e.g., candidiasis, coccidioidomycosis, cryptococcosis, cytomegalovirus disease, herpes simplex, lymphoma).
4. Autoimmune diseases requiring systemic immunosuppressive/immunomodulatory therapy within the past 2 years (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus).
5. Severe non-AIDS-related comorbidities, including uncontrolled clinically significant diseases of the genitourinary, cardiovascular, respiratory, neurological, psychiatric, gastrointestinal, endocrine, immune systems, or malignancies.
6. Central nervous system (CNS) disorders, such as epilepsy, cerebral ischemia/hemorrhage, dementia, cerebellar diseases, or autoimmune conditions involving the CNS.
7. Suspected or confirmed history of alcohol abuse, drug addiction, illicit substance use, or psychiatric disorders.
8. Abnormal laboratory results within 14 days prior to enrollment meeting any of the following:

   Hemoglobin <10 g/dL (female) or <11 g/dL (male) Absolute neutrophil count <1 ×10⁹/L Platelet count <100 ×10⁹/L Serum creatinine >110 μmol/L INR >1.5 or PTT >45 seconds ALT or AST >2.5 × upper limit of normal (ULN) Total bilirubin >1.5 × ULN
9. Current participation in another clinical trial that may conflict with the current protocol or outcome assessments.
10. Any other condition deemed inappropriate for participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-03-07 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions | Up to 12 Weeks After CAR T-cell Infusion

SECONDARY OUTCOMES:
HIV-1 RNA level | Up to 12 Weeks After CAR T-cell Infusion

OTHER OUTCOMES:
Immunological indicators | Up to 12 Weeks After CAR T-cell Infusion
CAR-T cell kinetics | Up to 12 Weeks After CAR T-cell Infusion

IPD SHARING:
Plan to Share IPD: No
We will share the results through published medical journal articles and at conference presentation after completion of the study.